CLINICAL TRIAL: NCT05007769
Title: A Phase II, Single-center, Open-label Study of Ramucirumab, Atezolizumab and N-803 After Progression on Any Immune Checkpoint Blocker in NSCLC (RAN)
Brief Title: Ramucirumab, Atezolizumab and N-803 After Progression on Any Immune Checkpoint Blocker in NSCLC
Acronym: RAN
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lost funding
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eli Lilly and Company (Industry); ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-x234
Record Dates: First submitted 2021-08-09; First posted 2021-08-16 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Non-small Cell Lung Cancer; Non-small Cell Carcinoma; NSCLC; Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Ramucirumab; atezolizumab; ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ramucirumab + Atezolizumab + N-803 (Experimental): -Ramucirumab intravenously (IV) on Day 1, atezolizumab IV on Day 1, and N-803 subcutaneous (SC) on Day 1 of each cycle. Cycles are 21 days.
  Interventions: Drug: Ramucirumab; Drug: Atezolizumab; Drug: N-803

INTERVENTIONS:
Drug: Ramucirumab — Will be supplied by Lilly Oncology, free of charge to the participant
  Other Names: Cyramza
Drug: Atezolizumab — Atezolizumab will be commercially available.
  Other Names: Tecentriq
Drug: N-803 — Will be supplied free of charge to the participants by ImmunityBio

SUMMARY:
The investigators hypothesize that the addition of ramucirumab and N-803 will augment the clinical activity of atezolizumab, and in order to evaluate the exact mechanism of action of the combination, the investigators propose a comprehensive analysis of paired peripheral blood samples collected during this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed squamous or non-squamous non-small cell lung cancer. Patients with known EGFR mutations, ALK or ROS1 rearrangements are not eligible.
* Availability of archival biopsy tissue or willingness to undergo a "baseline" biopsy prior to initiation of the trial for biomarker analysis, including PD-L1 by IHC. Results of the PD-L1 testing are not required for enrollment.
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan, as ≥ 20 mm by chest x-ray, or ≥ 10 mm with calipers by clinical exam.
* Prior use of an immune checkpoint blocker alone or in combination therapy. There is no limit on the number of lines of prior therapy a patient may have received.
* At least 18 years of age.
* ECOG performance status ≤ 1
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcl
  * Platelets ≥ 100,000/mcl
  * Hemoglobin ≥ 9.0 g/dL
  * Total bilirubin ≤ 1.5 x ULN
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x ULN or 5.0 x ULN in the setting of liver metastasis
  * Serum creatinine ≤ 1.5 x ULN or CrCl ≥ 40 mL/min. If serum creatinine is >1.5 times the ULN, a 24-hour urine collection to calculate creatinine clearance must be performed
* Adequate coagulation function as defined by:

  * INR ≤ 1.5
  * PTT/aPTT < 1.5 x ULN Note: Patients on full-dose anticoagulation must be on a stable dose of oral anticoagulant or low molecular weight heparin (LMWH) for a minimum duration of 28 days. If receiving warfarin, the patient must have an INR ≤3.0. For heparin and LMWH there should be no active bleeding (that is, no bleeding within 14 days prior to first dose of protocol therapy) or pathological condition present that carries a high risk of bleeding such as tumor involving major vessels or known varices.
* Urinary protein ≤ 1+ on dipstick or routine urinalysis. If urine dipstick or routine analysis is ≥ 2+, a 24-hour urine collection for protein must demonstrate < 1000 mg of protein in 24 hours to allow participation
* Because the teratogenicity of ramucirumab is not known, the patient, if sexually active, must be postmenopausal, surgically sterile, or using effective contraception (hormonal or barrier methods). Female patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to first dose of protocol therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study and for the duration of study participation.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

-Treatment with cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to Cycle 1, Day 1.

Note: Patients who have received acute, low-dose, systemic immunosuppressant medications such as one-time dose of dexamethasone for nausea or premedication for contrast dye allergy are eligible. The use of inhaled corticosteroids for chronic obstructive pulmonary disease (COPD) and fludrocortisone for patients with orthostatic hypotension or adrenocortical insufficiency is allowed. Patients using up to 10 mg of prednisone or equivalent per day are eligible.

* A history of other malignancy ≤ 3 years previous with the exception of patients with a negligible risk of metastasis or death and with expected curative outcome such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, or ductal carcinoma in situ treated surgically with curative intent or undergoing active surveillance per standard of care management including Rai Stage 0 chronic lymphocytic leukemia, prostate cancer with Gleason score ≤ 6 and prostate-specific antigen (PSA) ≤ 10 ng/mL.
* Having received any other investigational agents within 30 days or five times the half-life of the agent (whichever is sooner) of the planned start of the protocol therapy. Patients may be screened and consented but may not begin therapy within that 30 day washout period.
* Symptomatic or untreated asymptomatic brain metastases. Patients with treated brain metastases are eligible if they are clinically stable with regard to neurologic function, off steroids after cranial irradiation (whole brain radiation therapy, focal radiation therapy, and stereotactic radiosurgery) ending at least 2 weeks prior to randomization, or after surgical resection performed at least 28 days prior to randomization. The patient may have no evidence of Grade ≥1 CNS hemorrhage based on pretreatment MRI or IV contrast CT scan performed within 21 days before starting therapy.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to atezolizumab, ramucirumab, N-803, any other immune checkpoint blockade, chimeric or humanized antibodies, fusion proteins, or other agents used in the study.
* A history of prior severe immune-related adverse events requiring permanent discontinuation of the checkpoint inhibitors including all grade 4 toxicities and selected grade 3 toxicities such as pneumonitis, pancreatitis, neurological, cardiovascular, ocular, or renal adverse events.
* The patient is receiving chronic antiplatelet therapy, including dipyridamole or clopidogrel, or similar agents. Once-daily aspirin use (maximum dose 325mg/day) is permitted.
* The patient has experienced any arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 6 months prior to first dose of protocol therapy. Patients with unresected primary tumors or local recurrence who develop Grade 3 and 4 venous thromboembolism during the study may also receive anticoagulation and continue ramucirumab therapy provided that the tumor does not confer an excessive bleeding risk, in the opinion of the patient's physician.
* Uncontrolled or poorly controlled hypertension with blood pressure > 160 mmHg systolic or > 100 mmHg diastolic for > 4 weeks despite standard medical management.
* The patient has a prior history of GI perforation/fistula (within 6 months of first dose of protocol therapy) or risk factors for perforation.
* The patient has experienced any Grade 3 or 4 gastrointestinal bleeding within 3 months prior to first dose of protocol therapy.
* History of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis.
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug-induced), organizing pneumonia, or evidence of active pneumonitis on screening chest CT scan.
* Hemoptysis defined as bright red blood or ≥ ½ teaspoon within 2 months prior to Cycle 1 Day 1 or with radiographic evidence of intratumor cavitation or radiologically documented evidence of major blood vessel invasion or encasement by cancer.
* Serious or non-healing would, ulcer, or bone fracture within 28 days prior to Cycle 1 Day 1.
* Cirrhosis grade Child-Pugh B or C or cirrhosis of any degree with history of encephalopathy or clinically meaningful ascites, defined as requiring diuretics or paracentesis.
* Undergone major surgery within 28 days prior to Cycle 1 Day 1, minor surgery or subcutaneous venous access device placement within 7 days prior to Cycle 1 Day 1, or has elective or planned major surgery to be performed during the course of the clinical trial.
* Active tuberculosis.
* Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection with the former defined as HBV surface antigen (HBsAg) positive and HBV core antibody (HbcAb) positive with reflex positive HBV DNA. Note: Patients with past or resolved hepatitis B infection defined as having a negative HBsAg test and a positive HBcAb test or treated HCV with negative HCV RNA are eligible.
* Administration of a live, attenuated influenza vaccine within 4 weeks before Cycle 1 Day 1 or at any time during the study.
* Severe infections within 2 weeks prior to Cycle 1 Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia. Received oral or intravenous (IV) antibiotics within 2 weeks prior to Cycle 1 Day 1. Note: Patients receiving prophylactic antibiotics for prevention of a urinary tract infection or chronic obstructive pulmonary disease are eligible.
* History of deep venous thrombosis, pulmonary embolism, or any other significant thromboembolism during the 3 months prior to Cycle 1 Day 1. Venous port or catheter thrombosis or superficial venous thrombosis are not considered significant.
* Pregnant or breastfeeding. Women of childbearing potential must have a negative serum pregnancy test within 7 days of study entry.
* Known HIV-positivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-31 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Through completion of treatment (estimated to be 6 months)
  * ORR is defined as the proportion of participants achieving complete response or partial response measured according to RECIST 1.1
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

SECONDARY OUTCOMES:
Number of study treatment related adverse events as measured by NCI-CTCAE version 5.0 | From start of treatment through 30 days after completion of treatment (estimated to be 7 months)
Overall survival (OS) | Through completion of follow-up (estimated to be 30 months)
  -Defined as the duration of time from the start date of study treatment to death from any cause. Patients who are alive by the data cutoff date will be censored at the last follow up date.
Progression-free survival (PFS) | Through completion of follow-up (estimated to be 30 months)
  * PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  * Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Immune best overall response (iBOR) | Through completion of treatment (estimated to be 6 months)
  * Defined as the best time point response recorded from the start of the study treatment until the end of treatment, taking into account any requirement for confirmation.
  * iBOR will be measured by iRECIST criteria
Immune progression-free survival (iPFS) | Through completion of follow-up (estimated to be 30 months)
  * Defined by the first date at which progression criteria are met (i.e., the date of immune unconfirmed progression (iUPD) provided that immune confirmed progression (iCPD) is confirmed at the next assessment). If iUPD occurs, but later that patient develops immune stable disease (iSD), immune partial response (iPR), or immune complete response (iCR), then this initial iUPD date is not the date of PD. If progression is not confirmed and there is no subsequent iSD, iPR, or iCR, then the iUPD date should still be used in the following scenarios: if the patient stops protocol treatment because they were not judged to be clinically stable, or no further response assessments are done (because of patient refusal, protocol noncompliance, or patient death); the next time point response are all iUPD, and iCPD never occurs; or the patient dies from their cancer.
  * Progression will be measured per iRECIST criteria
Clinical benefit rate (CBR) | Through completion of treatment (estimated to be 6 months)
  * Defined as the percentage of participants who have achieved complete response, partial response, or stable disease measured according to RECIST 1.1
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Number of discontinuations due to treatment-related adverse events | From start of treatment through completion of treatment (estimated to be 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Morgensztern, M.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu